CLINICAL TRIAL: NCT07387497
Title: The Effect of Palm Stimulator Use During Peripheral Venous Catheterization on Pain, Fear, and Procedural Satisfaction in Cancer Patients Receiving Chemotherapy
Brief Title: Palm Stimulator Use During Peripheral Venous Catheterization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeliha CENGİZ (Other)
Responsible Party: Sponsor-Investigator, Zeliha CENGİZ, Associate Professor, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2026/9255
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Procedural Pain; Cancer; Fear Needles; Anxiety; Catheterization, Peripheral Venous
Keywords: Procedural Pain Management; Peripheral Venous Catheterization; Patient Satisfaction; Palm Stimulator; Oncology Nursing; Needle Fear; Tactile Stimulation
MeSH Terms: conditions — Pain, Procedural; Neoplasms; Iatrophobia; Anxiety Disorders; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Intervention Protocol: Participants will be randomized into two groups using Research Randomizer software:
  Palm Stimulator Group: 1-2 minutes before the procedure, patients will receive a brief orientation regarding the device. 20 seconds before PVC insertion, the device will be placed in the palm of the non-procedural hand. Patients will grip the device as the nurse applies the tourniquet. The tactile stimulation will continue throughout the needle entry and catheter stabilization.
  Control Group: Participants will receive the standard routine PVC protocol. No additional intervention will be provided during the procedure.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palm Stimulator Group (Experimental): 1-2 minutes before the procedure, patients will receive a brief orientation regarding the device. 20 seconds before PVC insertion, the device will be placed in the palm of the non-procedural hand. Patients will grip the device as the nurse applies the tourniquet. The tactile stimulation will continue throughout the needle entry and catheter stabilization.
  Interventions: Device: Palm Stimulator Group
- Control group (No Intervention): Participants will receive the standard routine PVC protocol. No additional intervention will be provided during the procedure.

INTERVENTIONS:
Device: Palm Stimulator Group — 1-2 minutes before the procedure, patients will receive a brief orientation regarding the device. 20 seconds before PVC insertion, the device will be placed in the palm of the non-procedural hand. Patients will grip the device as the nurse applies the tourniquet. The tactile stimulation will continue throughout the needle entry and catheter stabilization.
  Arms: Palm Stimulator Group

SUMMARY:
Purpose: The purpose of this study is to evaluate the effectiveness of a "Palm Stimulator" (a handheld device with blunt protrusions) in reducing pain, fear, and anxiety during peripheral venous catheterization (IV insertion) in adult cancer patients receiving chemotherapy.

Methods: This is a randomized controlled clinical trial. Participants will be randomly assigned to either the Experimental Group or the Control Group.

Experimental Group: During the IV insertion process, patients will hold and squeeze the Palm Stimulator in the palm of their non-procedural hand. The device is designed to provide intense tactile (touch) stimulation based on the "Gate Control Theory." Control Group: Patients will receive the standard routine care for IV insertion without any additional intervention.

Data Collection: Pain intensity will be measured using the Visual Analog Scale (VAS), while fear and anxiety levels will be assessed through VAS scales before and after the procedure. Patient satisfaction with the device will also be recorded.

Expected Outcome: The investigators hypothesize that the use of the Palm Stimulator will significantly decrease procedural pain and fear while increasing patient satisfaction compared to standard care. This study aims to provide a low-cost, non-pharmacological, and easy-to-use tool for oncology nurses to improve patient comfort during invasive procedures.

DETAILED DESCRIPTION:
Background: Cancer remains a complex disease that threatens individuals' lives across biopsychosocial dimensions. According to the World Health Organization, more than 19 million new cancer cases were diagnosed globally in 2020 (Sung et al., 2021). In modern oncology, chemotherapy is a primary treatment modality, with approximately 75% of these treatments administered intravenously (Duggan et al., 2024). Consequently, patients undergo repeated invasive procedures such as peripheral venous catheterization (PVC). Although PVC is a routine clinical task, it is a significant source of stress associated with pain, fear, and dissatisfaction. Inadequate management of procedural pain can lead to increased pain perception through peripheral and central sensitization, resulting in anticipatory anxiety and healthcare avoidance behaviors (Kapucu et al., 2017; Özırmak & Yayan, 2026).Oncology nurses bear critical responsibility in utilizing non-pharmacological methods to enhance patient comfort. Due to the side effects and cost limitations of pharmacological interventions, there is a need for low-cost, easy-to-integrate alternative approaches. While tactile stimulation-based interventions are promising, evidence regarding neurophysiologically based palmar stimulation is limited (Moustafa, 2024; Zengin & Yayan, 2022). The palm of the hand occupies a large representation area in the somatosensory cortex, allowing tactile stimuli from this region to be processed intensely by the central nervous system. Based on the Gate Control Theory, gripping the "Palm Stimulator" provides rapid sensory input that can inhibit pain perception at a neurophysiological level (Özırmak & Yayan, 2026).

Study Design and Setting: This study is designed as a randomized controlled clinical trial. It will be conducted at the Oncology Unit of Inönü University Turgut Ozal Medical Center between February and July 2026.

Intervention Protocol: Participants will be randomized into two groups using Research Randomizer software:

Palm Stimulator Group: 1-2 minutes before the procedure, patients will receive a brief orientation regarding the device. 20 seconds before PVC insertion, the device will be placed in the palm of the non-procedural hand. Patients will grip the device as the nurse applies the tourniquet. The tactile stimulation will continue throughout the needle entry and catheter stabilization.

Control Group: Participants will receive the standard routine PVC protocol. No additional intervention will be provided during the procedure.

Standardization: To ensure consistency, PVC procedures will be performed by nurses with at least one year of clinical experience. Standard 20G, 22G, or 24G catheters will be used. The Palm Stimulator (Utility Model No: 06479) will be disinfected with alcohol-based solutions between each use.

Data Collection and Tools: Data will be collected using face-to-face interviews and standardized scales:

Patient Identification Form: Demographic and clinical data (age, gender, diagnosis, chemotherapy cycle, etc.).

Visual Analog Scale (VAS): A 10 cm horizontal scale used to measure:Pre-procedural fear (0 = no fear, 10 = extreme fear).Post-procedural pain (0 = no pain, 10 = unbearable pain).Post-procedural satisfaction (0 = not satisfied, 10 = very satisfied).

Statistical Analysis:Data will be analyzed using IBM SPSS. Descriptive statistics (mean, SD, percentages) will be used for demographics. Normality will be tested via the Kolmogorov-Smirnov test. Independent Samples t-test or Mann-Whitney U test will be utilized for group comparisons. Pearson/Spearman correlation and ANCOVA will be performed to evaluate the relationship between pain scores and variables such as age or catheter size. The significance level is set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years.
* Receiving chemotherapy treatment via peripheral venous catheter (PVC).
* Cognitively capable of communicating and responding to pain, fear, and satisfaction scales.
* Volunteering to participate and providing written informed consent.

Exclusion Criteria:

* Diagnosis of chemotherapy-induced peripheral neuropathy or diabetic neuropathy.
* Presence of active infection, open wound, scar tissue, or edema in the palm.
* Use of analgesic medication within 4-6 hours before the procedure.
* History of hemiplegia or movement restriction in the extremity to be used for the procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Procedural Pain Intensity | Within 1 minute after the completion of the peripheral venous catheterization procedure.
  Procedural pain intensity will be measured using a 10-centimeter Visual Analog Scale (VAS), where 0 represents "no pain" and 10 represents "unbearable pain."

SECONDARY OUTCOMES:
Level of Procedural Fear | Immediately before the procedure and within 1 minute after the procedure.
  The level of fear regarding the injection will be assessed using the Visual Analog Scale (VAS-Fear), where 0 indicates "no fear" and 10 indicates "extreme fear." This assessment will be performed both before the procedure (pre-test) and after the procedure (post-test).
Patient Satisfaction With the Procedure | Within 1 minute after the completion of the procedure.
  Patients' satisfaction with the catheterization process and the intervention (if applicable) will be evaluated using a Visual Analog Scale (VAS-Satisfaction), where 0 represents "not satisfied at all" and 10 represents "very satisfied."

OTHER OUTCOMES:
Satisfaction With the Palm Stimulator | Within 5 minutes after the procedure.
  Patients in the intervention group will be asked two additional questions to evaluate their satisfaction specifically with the Palm Stimulator and their willingness to use it again in future procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Turgut Ozal Medical Center, Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with third parties or publicly to ensure the full protection of patient privacy and confidentiality, in accordance with the Law on the Protection of Personal Data (KVKK) and institutional ethical guidelines. The informed consent obtained from the participants does not include permission for the public sharing of raw individual data. Only de-identified, aggregated study results and statistical summaries will be presented through peer-reviewed publications and conference presentations to contribute to the scientific literature.

REFERENCES:
- [Background] Zengin M, Yayan EH. A Comparison of Two Different Tactile Stimulus Methods on Reducing Pain of Children During Intramuscular Injection: A Randomized Controlled Study. J Emerg Nurs. 2022 Mar;48(2):167-180. doi: 10.1016/j.jen.2021.10.006. Epub 2021 Dec 22. PMID 34952709
- [Background] Kapucu S, Ozkaraman AO, Uysal N, Bagcivan G, Seref FC, Eloz A. Knowledge Level on Administration of Chemotherapy through Peripheral and Central Venous Catheter among Oncology Nurses. Asia Pac J Oncol Nurs. 2017 Jan-Mar;4(1):61-68. doi: 10.4103/2347-5625.199081. PMID 28217732
- [Background] Duggan C, Hernon O, Dunne R, McInerney V, Walsh SR, Lowery A, McCarthy M, Carr PJ. Vascular access device type for systemic anti-cancer therapies in cancer patients: A scoping review. Crit Rev Oncol Hematol. 2024 Apr;196:104277. doi: 10.1016/j.critrevonc.2024.104277. Epub 2024 Mar 14. PMID 38492760
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Ozirmak N, Yayan EH. The difference between site of application and pain relief efficacy of the palm stimulator: A randomised controlled trial of intravenous blood drawn in children. J Pediatr Nurs. 2025 Nov 24;86:315-323. doi: 10.1016/j.pedn.2025.11.022. Online ahead of print. PMID 41289974